CLINICAL TRIAL: NCT03920150
Title: Vitamin D 24'000 IU for Oral Intermittent Supplementation
Acronym: DO-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00987
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Vitamin D Deficiency
Keywords: optimal vitamin D value
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Patient will be recruited by their general practitioner. Patients will be randomly assigned to be supplemented with monthly solution (control group), monthly capsules (IMP group) or weekly capsules after calculation of a individual loading dose (IMP + loading dose group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): 5 ml alcoholic solution containing 24'000 IU vitamin D for 3 months
  Interventions: Drug: Vitamin D3
- IMP (Active Comparator): Vitamin D oily capsules containing 24'000 IU vitamin D for 3 months
  Interventions: Drug: Vitamin D oily capsules
- IMP + loading dose (Active Comparator): Vitamin D oily capsules containing 24'000 IU vitamin D for an individual number of weeks calculated with the formula: 40 x (100 - actual value [nmol/l] x body weight [kg] / 24'000 IU.
  Interventions: Drug: Vitamin D oily capsules

INTERVENTIONS:
Drug: Vitamin D3 — Patient will be treated with 3 doses of alcoholic solution for 3 months.
  Other Names: Vi-De 3 Monatsdosis
  Arms: Control
Drug: Vitamin D oily capsules — Patient will be treated with 3 capsules for 3 months.
  Arms: IMP
Drug: Vitamin D oily capsules — Patient will be treated with weekly capsules for an individually calculated number of weeks.
  Arms: IMP + loading dose

SUMMARY:
Vitamin D deficiency (defined as 25(OH)-vitamin D serum level <50 nmol/l) is cured with oral supplementation. National guidelines recommend the administration of 800 IU cholecalciferol daily for an effective treatment, especially during the winter (poor sun exposition). Cumulative intermittent administration monthly (24'000 IU) or weekly (5'600 IU) is possible. Commercially available intermittent pharmaceutical forms in Switzerland are liquid (oily or alcoholic solution). The study aims to compare the rise of vitamin D3 levels after treatment between newly developed soft capsules and monthly solution (primary outcome), and to evaluate the effect of a loading dose (without infringing the cumulative maximal dose of 4'000 IU per day) on the achievement of optimal values >75 nmol/l (secondary outcome). The investigators will use newly developed soft capsules and alcoholic solution, which are commercially available in Switzerland.

DETAILED DESCRIPTION:
Group Control, Alcoholic Drinking Solution: 5 ml of an alcoholic drinking solution with 24'000 IU vitamin D p.o. once a month for 3 months (3 doses).

Group IMP, Capsules: one capsule with 24'000 IU vitamin D p.o. once a month for 3 months (3 doses).

Group IMP + loading dose, Loading Dose: one capsule with 24'000 IU vitamin D p.o. once a week during an individually calculated number of weeks.

All 3 groups: Measurement of vitamin D in serum before therapy and one week after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* vitamin D deficiency by serum level <50 nmol/l

Exclusion Criteria:

* hypercalcaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Serum level of vitamin D | 3 months of treatment
  Level of serum vitamin D after 3 month treatment compared to baseline value

SECONDARY OUTCOMES:
Serum level of vitamin D after loading dose | up to 4 months of treatment
  Level of serum vitamin D > 75 nmol/l after an individual number of treatment weeks, calculated with a loading dose formula.
Adverse Drug Reactions | 3 months of treatment
  Number and severity of adverse drug reactions during treatment
Adherence to medication | 3 months of treatment
  Taking adherence: (number of doses taken) divided by (number of doses prescribed) x 100.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof, Study Chair — Pharmaceutical Care Research Group
Locations (1):
- Pharmaceutical Care Research Group, Basel, Switzerland